CLINICAL TRIAL: NCT07252219
Title: Effects of Ankle Evertor Fatigue on Force Sense and Neuromuscular Activation During Submaximal Isometric Contractions in Individuals With and Without Chronic Ankle Instability
Brief Title: Effects of Ankle Evertor Fatigue on Force Sense and Neuromuscular Activation in Subjects With Chronic Ankle Instability
Status: Recruiting | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Alan Kacin, Head of Laboratory, University of Ljubljana
Other Study IDs: 0120-197/2023/3/isokinetic
Record Dates: First submitted 2025-09-10; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: chronic ankle instability; force sense; muscle fatigue; proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Healthy participants without a history of ankle sprain or self-reported ankle instability. Participants will complete the same experimental protocol as the group of chronic ankle instability, including a fatigue protocol of the ankle evertors
- Chronic ankle instability group: Participants with chronic ankle instability, defined by a history of recurrent ankle sprains and self-reported instability. Participants will complete the same experimental protocol as the control group, including a fatigue protocol of the ankle evertors.

SUMMARY:
The goal of this observational study is to investigate whether ankle evertor muscle fatigue impairs force perception and alters neuromuscular activation patterns during submaximal isometric contractions, and whether these effects differ between individuals with chronic ankle instability (CAI) and individuals without CAI.

DETAILED DESCRIPTION:
Participants will first be familiarized with the research protocol for approximately 20 minutes. After a short break, the experimental protocol with data collection will begin and last between 45 and 60 minutes. Measurements will be performed on the side where the participant reports symptoms of chronic ankle instability. In cases of bilateral CAI, the leg with the lower CAIT score will be tested.

Participants will be tested on an isokinetic dynamometer (Humac Norm, CSMi, USA) in a semi-recumbent position with the hip and knee flexed to ensure comfort and alignment. The trunk and tested leg will be secured with straps to minimize accessory movement. After initial maximal voluntary isometric contraction (MVIC) of ankle evertors, participants will perform force-matching tasks at 25% and 50% of MVIC. Each trial will consist of 5 seconds with visual feedback followed by 5 seconds without feedback, repeated three times per intensity. After completing these tasks, participants will undergo a fatigue protocol for the ankle evertors. After the fatigue protocol, participants will repeat the force-matching tasks at both 25% and 50% MVIC.

The muscle fatigue protocol consists of consecutive isotonic contractions of ankle eversion, performed through the full range of motion at 30% of MVIC torque until visible fatigue. Fatigue will be defined as a clear inability to perform full range of eversion, i.e. the range of motion fell below 10% of the initial value despite evident effort by the participant. The test will be paced using a metronome, with a 1-second concentric and a 1-second eccentric phase to ensure consistent movement velocity.

ELIGIBILITY:
Inclusion criteria for the healthy control group (no CAI):

* Age between 18 and 45 years,
* No history of injuries or surgical procedures to the lower limbs,
* No peripheral or central neurological impairments.

Inclusion criteria for the chronic ankle instability (CAI) group:

* Age between 18 and 45 years,
* No history of major surgical procedures on the lower limbs
* No peripheral or central neurological impairments,
* Diagnosed chronic ankle instability:

  * First ankle sprain occurred at least one year prior to testing,
  * At least three months since the most recent ankle sprain,
  * Subjective feeling of ankle instability - CAIT (Cumberland Ankle Instability Tool) score < 24.

Exclusion criteria for the CAI group:

- Other pathologies of the ankle joint.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited by convenience sampling from the general population and clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Constant Error (CE) | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Muscle force sense will be assessed by the accuracy of force reproduction during force-matching tasks.
  Constant Error (CE) will be calculated as the mean difference in force (Nm) between reproduction with and without visual feedback during the middle three seconds, averaged across three repetitions at each load level.
  Unit of measure: Newton-meters (Nm).
Absolute Error (AE) | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Muscle force sense will be assessed by the accuracy of force reproduction during force-matching tasks.
  Absolute Error (AE) will be calculated as the mean absolute difference in force (Nm) between reproduction with and without visual feedback during the middle three seconds, averaged across three repetitions at each load level.
  Unit of measure: Newton-meters (Nm).
Variable Error (VE) | Time Frame: Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Muscle force sense will be assessed by the accuracy of force reproduction during force-matching tasks.
  Variable Error (VE) will be calculated as the standard deviation of errors across three repetitions at each load level.
  Unit of measure: Newton-meters (Nm).
Coefficient of Variation (CV) of generated force | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Ratio of the standard deviation to the mean force during the middle three seconds of sustained contraction in each trial, calculated separately for trials with and without visual feedback. Unit of Measure: Percentage (%).

SECONDARY OUTCOMES:
Surface EMG root mean square (RMS) amplitude of ankle muscles | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  RMS amplitude from surface EMG signals of the peroneus longus, tibialis anterior, soleus, and gastrocnemius medialis will be obtained during the fatigue protocol, MVIC and force-matching task. Unit of Measure: millivolts (mV).
Surface EMG median frequency of peroneus longus mucle | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Median frequency of EMG signals will be obtained from the peroneus longus during the fatigue protocol, the maximal voluntary isometric contraction (MVIC) and force-matching tasks. Frequency values will be averaged across repetitions. Unit of Measure: Hertz (Hz).
Maximal voluntary isometric contraction (MVIC) | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  MVIC of the ankle evertors will be measured at the beginning of the protocol to determine the target force for submaximal isometric contractions, and repeated immediately after the fatigue protocol to assess the effectiveness of fatigue, expressed in Newton-meters (Nm).
Ratings of perceived exertion | Baseline (Day 1, prior to fatigue protocol) and immediately post-fatigue (Day 1, within 5 minutes after fatigue protocol).
  Description: Ratings of perceived exertion (RPE) will be assessed at the end of each fatigue protocol using the Borg 10 category-ratio scale, with 0 is no effort and 10 is an extreme physical effort.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD in anonymized form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No limit.
Access Criteria: All IPD will be shared upon reasoned request for the purpose of further scientific analysis (i.e. systematic reviews, meta-analyzes, etc.). A proposal describing the planned analyzes must be submitted in writing to the principal investigator, Dr. Alan Kacin, by email to alan.kacin@zf.uni-lj.si.